CLINICAL TRIAL: NCT06993506
Title: Sacituzumab Tirumotecan Monotherapy or Combination Therapy in Patients With Unresectable Locally Advanced, Recurrent or Metastatic HER2-Negative Breast Cancer: A Real-World Study
Brief Title: Real-world Study of SKB264 Monotherapy or Combination Therapy in Recurrent or Metastatic HER2-negative Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, PENG YUAN, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC5312
Record Dates: First submitted 2025-05-12; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: HER2-negative Breast Cancer; Recurrence; Metastasis
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis | interventions — Combined Modality Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TNBC Cohort: * Histological/cytological confirmed of triple-negative breast cancer (TNBC) from the most recent pre-SKB264 biopsy/pathological report, with: HER2 negative: immunohistochemistry (IHC) of 0 or 1+; if is 2+ by IHC, negative HER2 expression must be confirmed by fluorescence in situ hybridization (FISH); Estrogen and progesterone receptor negative means that less than 1% of the cells express hormone receptors as indicated by IHC;
  * Locally advanced, recurrent, or metastatic disease (locally advanced disease should be confirmed by investigators as ineligible for curative resection)
  Interventions: Drug: SKB264 Monotherapy or Combination Therapy
- HR+/HER2- BC Cohort: * Histological/cytological confirmed of HR+/HER2- breast cancer from the most recent pre-SKB264 biopsy/pathological report, with: HER2 negative: IHC of 0 or 1+; if is 2+ by IHC, negative HER2 expression must be confirmed by FISH; HR positive: Hormone receptor-positive (HR, ER, or PR status) was defined as ≥1% expression by IHC.
  * Locally advanced, recurrent, or metastatic disease (locally advanced disease should be confirmed by investigators as ineligible for curative resection);
  Interventions: Drug: SKB264 Monotherapy or Combination Therapy

INTERVENTIONS:
Drug: SKB264 Monotherapy or Combination Therapy — The interventions in this study comprised SKB264 monotherapy or combination therapy involving SKB264. The specific combination regimens were determined based on real-world clinical practice.

SUMMARY:
This study is a multi-center observational real-world study, with a total of 500 patients planned to be enrolled. This study is divided into two cohorts: the triple-negative breast cancer (TNBC) cohort and the hormone receptor-positive/human epidermal growth factor receptor 2-negative breast cancer (HR+/ HER2-BC) cohort. The aim of this study is to assess the efficacy and safety of Sacituzumab Tirumotecan (SKB264) monotherapy or combination therapy in patients with unresectable locally advanced, recurrent or metastatic HER2-negative breast cancer in the real-world setting.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years old at the time of signing the informed consent form, regardless of gender;
2. Patient must meet one of the following pathological diagnoses and classifications:

   2.1) For TNBC Cohort: -Histological/cytological confirmed of triple-negative breast cancer (TNBC) from the most recent pre-SKB264 biopsy/pathological report, with: HER2 negative: immunohistochemistry (IHC) of 0 or 1+; if is 2+ by IHC, negative HER2 expression must be confirmed by fluorescence in situ hybridization (FISH); Estrogen and progesterone receptor negative means that less than 1% of the cells express hormone receptors as indicated by IHC; -Locally advanced, recurrent, or metastatic disease (locally advanced disease should be confirmed by investigators as ineligible for curative resection); 2.2) For HR+/HER2- BC Cohort: -Histological/cytological confirmed of HR+/HER2- breast cancer from the most recent pre-SKB264 biopsy/pathological report, with: HER2 negative: IHC of 0 or 1+; if is 2+ by IHC, negative HER2 expression must be confirmed by FISH; HR positive: Hormone receptor-positive (HR, ER, or PR status) was defined as ≥1% expression by IHC.-Locally advanced, recurrent, or metastatic disease (locally advanced disease should be confirmed by investigators as ineligible for curative resection);
3. Plan to receive SKB264 monotherapy or combination therapy;
4. Prior treatment lines: -For TNBC Cohort: ≤2 lines of systemic antitumor therapy for unresectable locally advanced, recurrent, or metastatic disease; -For HR+/HER2- BC Cohort: ≤2 lines of systemic antitumor therapy (excluding endocrine therapy) for unresectable locally advanced, recurrent, or metastatic disease;
5. Voluntarily participate in the study, sign the informed consent form and demonstrate good compliance.

Exclusion Criteria:

1. Patients with other malignancies, except cured basal or squamous cell skin cancer or in situ cancer of cervix; and patients with other malignancies must have a tumor-free period of at least 5 years;
2. Patients who are currently participating in other interventional clinical studies;
3. Known allergy to the investigational drug or any of its components;
4. Pregnant or lactating women;
5. Any situation that the researchers consider to interfere with the evaluation of the study drug or the safety of the subjects or the analysis of the study results, or any other situation that the researchers consider inappropriate to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Unresectable Locally Advanced, Recurrent or Metastatic HER2-Negative Breast Cancer
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Time to next treatment (TTNT) of SKB264 monotherapy or combination therapy in patients with unresectable locally advanced, recurrent or metastatic HER2-negative breast cancer | Time from initiation of SKB264 monotherapy or combination therapy to start of next treatment, assessed up to 24 weeks.

SECONDARY OUTCOMES:
Real world progression free survival (rwPFS) of SKB264 monotherapy or combination therapy | Time from initiation of SKB264 monotherapy or combination therapy to the first documented evidence of progression or death, whichever came first, assessed up to 24 weeks.
Duration of treatment (DOT) of SKB264 monotherapy or combination therapy | Time from initiation of SKB264 monotherapy or combination therapy to its discontinuation, assessed up to 24 weeks.
Real world objective response rate (rwORR) of SKB264 monotherapy or combination therapy | The proportion of patients who had a complete or partial response documented by imaging reports or by assessment of treating physician during the study treatment, which is approximately up to 24 weeks from the initiation of the study treatment.
Real world overall survival (rwOS) of SKB264 monotherapy or combination therapy | Time from initiation of SKB264 monotherapy or combination therapy to death from any cause, assessed up to 48 weeks.
Number of patients with adverse events of SKB264 monotherapy or combination therapy in the real-world setting, graded and recorded according to NCI CTCAE v5.0. | Adverse events were assessed during study treatment and at follow-up visits, which is approximately up to 30 weeks from the initiation of the study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No